CLINICAL TRIAL: NCT00986700
Title: The Effect of Late Night Meals on Fasting Glucose in Type 2 Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Jacob Ilany MD, Senior Endocrinologist, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-09-7156-JI-CTIL
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Fasting Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- different types of bad time food (Other): Different types of bad time food
  Interventions: Dietary Supplement: late night meal

INTERVENTIONS:
Dietary Supplement: late night meal — Three different kinds of late night meal each for 2 days.

SUMMARY:
High fasting glucose is a very common problem in type 2 diabetic patients. The cause is probably glucose production by the liver, known as the "dawn phenomenon". The investigators hypothesize that a late night meal can lower the fasting glucose level by early morning insulin secretion stimulated by the food. In this study the investigators intend to test the effect of different kinds of late night meals on fasting glucose in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus with HbA1c 6.5-9%, fasting glucose of 126-200 mg/dl and BMI of 27-40.

Exclusion Criteria:

* Patient treated with insulin, GLP-1 analog or weight reduction medications.
* Type 1 diabetes
* Pregnancy
* Renal failure (creatinin >1.4 for male and 1.3 for female
* Uncontrolled hypertension (>160/100)
* Abnormal thyroid function test
* Patient treated with steroids or psychiatric medications.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
fasting glucose level | 2 weeks